CLINICAL TRIAL: NCT02736500
Title: Peptide Receptor Radionuclide Therapy With 177Lu-Dotatate Associated With Metronomic Capecitabine In Patients Affected By Aggressive Gastro-Etero-Pancreatic Neuroendocrine Tumors
Acronym: LuX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Istituto Europeo di Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.19
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors; Gastro Entero Pancreatic Neuroendocrine Tumors
Keywords: neuroendocrine tumors; gastro entero pancreatic neuroendocrine tumors; Radioisotope therapy; 177Lu-DOTATATE; METRONOMIC CAPECITABINE
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 28 GBq 177Lu-DOTATATE (Experimental): 5 cycles of 5.5 GBq (150 mCi) each, up to the total cumulative activity of 28 GBq (750 mCi) 177Lu-DOTATATE
  Interventions: Drug: 28 GBq 177Lu-DOTATATE
- 22 GBq 177Lu-DOTATATE (Experimental): 6 cycles of 3.7 GBq (100 mCi) each, up to the total cumulative activity of 22 GBq (600 mCi) 177Lu-DOTATATE
  Interventions: Drug: 22 GBq 177Lu-DOTATATE

INTERVENTIONS:
Drug: 28 GBq 177Lu-DOTATATE — Patients without risk factors (particularly long standing and poorly controlled diabetes and hypertension) for late renal toxicity will be administered with 5 cycles of 5.5 GBq (150 mCi) each, up to the total cumulative activity of 28 GBq (750 mCi) of 177Lu-DOTATATE.
  Arms: 28 GBq 177Lu-DOTATATE
Drug: 22 GBq 177Lu-DOTATATE — Patients with risk factors for late renal toxicity will be administered with 6 cycles of 3.7 GBq (100 mCi) each, up to the total cumulative activity of 22 GBq (600 mCi)177Lu-DOTATATE
  Arms: 22 GBq 177Lu-DOTATATE

SUMMARY:
The aim of this phase I-II study is to evaluate the efficacy and toxicity of PRRT with 177Lu-DOTATATE (Lu-PRRT) associated to metronomic chemotherapy with Capecitabine in patients affected by aggressive FDG-positive gastro-entero-pancreatic NET. Moreover to analyze the effects of the capecitabine metronomic schedule on the level of circulating angiogenetic factors.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are relatively rare tumors, mainly originating from the digestive system, able to produce bioactive amines and hormones. NETs tend to be slow growing and are often diagnosed when metastatic. Treatment is multidisciplinary and should be individualized according to the tumor type, burden, and symptoms. Therapeutic tools include surgery, interventional radiology, and medical treatments such as somatostatin analogues, interferon, chemotherapy, new targeted drugs (everolimus, sunitinib) with radiolabelled somatostatin analogues. Despite the options available, antiproliferative treatment options for patients with inoperable gastro-entero-pancreatic (GEP) NETs are limited.

PRRT with radiolabelled somatostatin analogues 90Y-DOTATOC, and 177Lu-DOTATATE (177Lu-DOTA-D-Phe1-Tyr3-octreotate), has been experimented for more then 15 years in few centers. The introduction of PRRT and, particularly, the advent of 177Lu-DOTATATE, broke through the poor scenario of available treatment for NETs.

Dosimetric studies demonstrated that 90Y-DOTATOC and 177Lu-DOTATATE are able to deliver high radiation doses to somatostatin receptor sst2-expressing tumors and low doses to normal organs. Clinical studies demonstrated that partial and complete objective responses in up to 30% of patients can be obtained, with a great survival benefit including those with stable disease. Side effects may involve the kidney and the bone marrow and are usually mild. Renal protection is used to minimize the risk of a late decrease of renal function.

Recently, in order to further increase the objective response to PRRT, a combined treatment with the radiosensitizer capecitabine, has been proposed and tested on GEP-NET patients' population. Capecitabine is the oral prodrug of 5-fluorouracile (5-FU), which is active in GEP tumors and a radiosensitizer itself. The finding that neo-angiogenesis can be shut down also with cytotoxic drugs like capecitabine when administered in low and frequent doses, constitutes the rationale for proposing a particular schedule of chemotherapy that is, therefore, named "metronomic" or "anti-angiogenic".

Based on the reported experience, the investigators think to offer a combined therapy in aggressive, metabolically active tumors, such as those patients with a positive FDG scan. FDG-PET allow the investigators to obtain in vivo imaging of increased glycolysis which is known to be an hallmark of tumor aggressiveness.

The aim of this phase I-II study is to evaluate the efficacy and toxicity of PRRT with 177Lu-DOTATATE (Lu-PRRT) associated to metronomic chemotherapy with Capecitabine in patients affected by aggressive FDG-positive gastro-entero-pancreatic NET. Moreover to analyze the effects of the capecitabine metronomic schedule on the level of circulating angiogenetic factors.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic diagnosis of inoperable or metastatic gastro-entero-pancreatic neuroendocrine neoplasia.
* Conserved hematological, liver and renal parameters: haemoglobin >= 10 g/dL, absolute neutrophil count (ANC) >= 1.5 x 109 /L, platelets >= 100 x 109 /L, bilirubin ≤1.5 X UNL (upper normal limit), ALT <2.5 X UNL (< 5 X UNL in presence of liver metastases), creatinine < 2 mg/dL.
* Age more than 18 years.
* Patients with documented disease will be admitted to therapeutic phase only if the diagnostic receptor imaging (OctreoScan) demonstrate a significant uptake in the tumor (grade 2 or 3, according to a preset scoring, where grade 1= equal to normal liver, grade2 = higher than normal liver, grade 3= higher than kidneys and spleen), that may allow delivering a low absorbed dose to normal organs and a high dose to the tumor.
* Patients with documented disease will be admitted to therapeutic phase only if the 18FDG PET/CT is positive with a SUV > 2.5 at least in one documented lesion.
* Disease must be measurable by means of conventional imaging (CT or MRI).
* Before treatment clinical history data will be collected, physical examination will be performed and diagnostic and laboratory data will be examined.
* Patients must not receive other treatments (e.g. chemo- or radiotherapy) from one month before to two months after the completion of 177Lu-DOTATATE cycles.
* Patients must be naive from previous radionuclide treatments with radiopeptides (e.g. 111Inpentetreotide, 90Y-DOTATOC) or other radiopharmaceuticals (e.s. 131I-MIBG, 131I).

Exclusion Criteria:

* Pregnancy/breastfeeding (a pregnancy test not older than 7 days is mandatory).
* Assessed bone marrow invasion > 25%.
* Other concomitant neoplasm (excluding in situ basaliomas and radically treated cervical cancers).
* ECOG score higher than 2.
* Expectancy of life shorter than 6 months.
* Patients with psycho-physical conditions that are not suitable for entering this clinical study and fulfilling its requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Objective Overall Response Rate | up to 24 months
  rate of objective clinical response (complete response (CR), partial response (PR), or minor response (MR) according to RECIST criteria
toxicity rate | up to 24 months
  The rate of toxicity, either acute or delayed, according to NCI criteria, of the association 177Lu-DOTATATE and metronomic capecitabine.

SECONDARY OUTCOMES:
Progression free survival in association with histopathology characteristics | up to 24 months
  evaluation of the PFS and the possible association between histopathology characteristics (grading and proliferation index)
Progression free survival in association with the receptor and metabolic status at OctreoScan and FDG PET | up to 24 months
  Progression free survival in association with the receptor and metabolic status at OctreoScan and FDG PET

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Paganelli, MD, Principal Investigator — IRST IRCCS, Meldola (FC)
Locations (2):
- Italy (2):
  - Giovanni Paganelli, Meldola, FC
  - Lisa Bodei, Milan